CLINICAL TRIAL: NCT03316222
Title: Phase 1/2a Study to Evaluate the Safety, Activity, and Pharmacokinetics of Escalating Doses of GNS561 in Patients With Primary and Secondary Liver Cancer
Brief Title: Study of GNS561 in Patients With Liver Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: only phase 1b was completed and the phase 2 will be an another study, finally
Sponsor: Genoscience Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNS561-CL-I-Q-0211
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma, Intrahepatic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Dose escalation using 3+3 design with dose limiting toxicity (DLT) observation period of 28 days.
  Interventions: Drug: GNS561
- Dose Expansion (Experimental): Additional patients will be enrolled into the recommended dose. These additional patients will undergo all of the same assessments as the patients enrolled in dose escalation with the exception of PK sampling.
  Interventions: Drug: GNS561

INTERVENTIONS:
Drug: GNS561 — Escalating doses to be administered 3 times a week.

SUMMARY:
This is a first in human, open-label dose escalation study to investigate the safety, tolerability and pharmacokinetics of GNS561 in patients Primary and Secondary liver cancer

DETAILED DESCRIPTION:
This is a multicenter, open-label, uncontrolled, repeat-dose Phase 1/2a study designed to evaluate the safety profile and to determine the recommended Phase 2 dose of GNS561 in patients with advanced primary and secondary liver cancer. This study will enroll approximately 50 patients and consists of 2 parts: Phase 1(dose escalation) and Phase 2 (expansion). All patients will be treated until the occurrence of an unacceptable toxicity, disease progression, or withdrawal of consent. In this study a treatment cycle is defined as 4 weeks (28 days). Patients are to take their assigned dose of GNS561, in the Morning and in the evening at the same time everyday, following a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Histologically confirmed and documented locally advanced or metastatic HCC that is deemed not appropriate for curative therapy and Histologically confirmed and documented locally advanced or metastatic iCCA.
3. Liver tumor burden< 50% of the liver (per Investigator judgment)
4. Antiviral therapy required in hepatitis B virus patients (Hepatitis B antigen positive)
5. Willing to have liver biopsy at the beginning of cycle 2 (Day 1)
6. Presence of a measurable tumor per RECIST v1.1 criteria
7. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
8. Life expectancy ≥ 12 weeks
9. Adequate hematologic function prior to the first dose of GNS561, defined as:

   1. Absolute neutrophils count ≥ 1500 cells/µL
   2. Hemoglobin ≥ 10 g/dL with no transfusion within 4 weeks prior to first planned dose of GNS561
   3. Platelet count > 50,000/µL with no transfusion within 2 weeks prior to first planned dose of GNS561
10. Adequate renal function prior to first dose, defined as

    1. Serum creatinine < 1.5 ULN
    2. Creatinine clearance ≥ 50 mL/min/m2 (by Cockroft-Gault equation of 24-hour urine) if creatinine ≥ 1.5 X ULN
11. Adequate hepatic function prior to first dose, defined as AST/ALT ≤ 5 X ULN
12. Women patients of childbearing potential must have a negative serum/urine pregnancy test at screening and baseline, and be willing to use a medically acceptable form, as judged by Investigator and Sponsor, of contraception (e.g., hormonal birth control, intrauterine device [IUD], or barrier method [male condom, female condom, diaphragm]), plus a spermicidal agent [contraceptive foam, jelly, or cream]) or abstinence or bilateral occlusion or whose partner had a vasectomy at least 2 years before screening. The patient should be advised to continue the contraception for at least 6 months following the completion of dosing. Women with cessation for > 24 months of previously occurring menses, or women of any age who have had a hysterectomy, or have had both ovaries removed will be considered to be of non-childbearing potential.
13. Male patients of reproductive potential must be willing to use one acceptable method of contraception, as judged by Investigator and Sponsor, as described in Criteria 12 and/or to refrain from donating sperm from the time of screening through at least 6 months following the completion of dose administration.
14. Amenable to computed tomography (CT) with 3 or 4 phase liver or magnetic resonance imaging (MRI) of abdomen and pelvis, and CT of chest, or MRI of whole body, for initial tumor size measurements and subsequent follow-up.
15. Absence of other clinically relevant abnormalities for screening laboratory test results as judged by the Investigator and Sponsor.
16. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
17. Be willing to abstain from alcohol from signing of informed consent through Week 5 (completion of PK sampling at the beginning of Cycle 2).
18. Able to understand and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding mothers
2. Any known history of encephalopathy
3. Known esophageal varices with recent history of bleeding (within previous 2 months)
4. Clinically significant ascites or paracentesis
5. Known untreated or symptomatic brain metastases
6. Presence of residual toxicities of ≥ Grade 2 after prior antitumor therapy ≤ 4 weeks prior to first dose. Grade 1 toxicities related to previous treatments are acceptable at the time of the first planned dose of GNS561, as well as any alopecia.
7. Chronic treatment with immunosuppressive agents (like steroids) ≤ 6 weeks prior to first planned dose of GNS561.
8. Major surgical procedures, open biopsy or significant traumatic injury ≤ 4 weeks prior to first dose of GNS561 or anticipation of major surgical procedure during the course of the trial, minor surgical procedures ≤ 1 week of first planned dose
9. Any clinically significant cardiovascular condition as judged by the Investigator
10. Severe or uncontrolled renal condition
11. Untreated chronic hepatitis B
12. Known history of immunodeficiency diseases (e.g., active HIV)
13. Use of any prohibited concomitant medications within 14 days of the Baseline/Day 1 visit
14. Known current alcohol (> 20g/ Day in women and > 30g/ Day in men) or substance abuse
15. Malabsorption issues (e.g., gastric bypass or gastrectomy patients)
16. Participation in any investigational clinical investigation ≤ 4 weeks prior to first planned dose of GNS561 or longer if required by local regulations, and for any other limitation of participation based on local regulations
17. Known clinically significant or life threatening organ or systemic disease such that in the opinion of the Investigator, the significance of the disease will compromise the patient's participation in the trial
18. Is a participant or plans to participate in another investigational clinical study, while taking part in this study.
19. Known intolerance or hypersensitivity to the active ingredient or to one of the components of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | Dose-Limiting Toxicity will be evaluated during the 4 - week dose escalation phase.
  Dose-Limiting Toxicity will be measured by adverse events by dose level

CONTACTS AND LOCATIONS:
Locations (5):
- Memorial Sloan Kettering, New York, New York, United States
- Jules Bordet Institute, Brussels, Belgium
- France (3):
  - CHU Grenoble, Grenoble
  - Croix-Rousse Hospital, Lyon
  - Saint-Joseph Hospital, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harding JJ, Awada A, Roth G, Decaens T, Merle P, Kotecki N, Dreyer C, Ansaldi C, Rachid M, Mezouar S, Menut A, Bestion EN, Paradis V, Halfon P, Abou-Alfa GK, Raymond E. First-In-Human Effects of PPT1 Inhibition Using the Oral Treatment with GNS561/Ezurpimtrostat in Patients with Primary and Secondary Liver Cancers. Liver Cancer. 2022 Feb 15;11(3):268-277. doi: 10.1159/000522418. eCollection 2022 Jun. PMID 35949290